CLINICAL TRIAL: NCT00680927
Title: Reveal® XT Performance Trial
Brief Title: Reveal® XT Performance Trial (XPECT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Responsible Party: Medtronic Bakken Research Center BV, Medtronic Bakken Research Center BV
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CMD 446
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2009-01

CONDITIONS: Atrial Fibrillation; Risk of Cardiac Arrhythmias
Keywords: Atrial Fibrillation; Risk of cardiac arrhythmias; Loop recorder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: 46 hrs Holter ECG recording — Maximum of 2 46 hrs external Holter ECG recordings are required.

SUMMARY:
The purpose of this study is to quantify the accuracy of the atrial fibrillation diagnostics of the Reveal® XT in a clinical setting and to verify overall system performance, R-wave sensing performance, to obtain user feedback, from both patient and physician, and collect data on device safety.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, multi-center international post-market study.

The study will be conducted at 20-30 centers primarily in Europe. The study will be conducted at least in Germany, Austria, Switzerland, The Netherlands, and the Czech Republic. Study centers from Canada may also participate, depending on the timelines for regulatory approval and commercial release of the Reveal® XT in this region.

It is expected that between 140 and 200 patients will be enrolled to ensure that at least 47 patients are included to assess the first primary objective and at least 60 patients to assess the second primary objective.

The primary objective is to quantify the AF detection performance of the device.

The patient population will be assessed in two separate cohorts. The first primary objective is to quantify the 24-hour AF burden accuracy in patients with more than 1% AF burden.

The second primary objective is to quantify the detection accuracy of non-arrhythmia in patients with 1% or less AF burden.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to provide his/her informed consent
* Patient has been implanted with a Reveal® XT
* Patient fulfills at least one of the following three additional requirements

  1. is scheduled for PV ablation or surgical rhythm control intervention, and the PV ablation or surgical intervention can be deferred until study completion or
  2. has documented frequent AF or frequent symptoms attributable to AF or
  3. has undergone PV ablation within the last 6 months and still has symptoms attributable to AF

Exclusion Criteria:

* Patient has an implanted pacemaker or ICD
* Patient has persistent or permanent AF
* Patient is allergic to adhesive ECG electrodes
* The study will interfere with a therapeutic or diagnostic procedure which is planned or expected during the study period
* Patient is participating in another study that is expected to compromise the results of this study
* Patient is a minor, legally incompetent, or does not meet other local requirements for participation in a clinical study
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation Burden (AF Burden) | 46 hrs

SECONDARY OUTCOMES:
AF episode detection accuracy and AF episode duration accuracy | 46 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Guido H. Rieger, MD, Study Director — Medtronic Bakken Research Center B.V.; Gerhard Hindricks, MD, PhD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (24):
- Austria (3):
  - LKH - Universitätskliniken, Innsbruck
  - A.ö. Krankenhaus der Elisabethinen Linz, Linz
  - Salzburger Landeskliniken, Salzburg
- University Gasthuisberg, Leuven, Belgium
- Canada (3):
  - Hopital Laval, Québec
  - St. Paul's Hospital, Vancouver
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria
- Czechia (3):
  - Facultni Nemocnice Brno, Brno
  - Nemocnice Na Homolce Hospital, Prague
  - Klinika Kardiologie IKEM, Prague
- Germany (7):
  - Herzzentrum Bad Krozingen, Elektrophysiologie, Bad Krozingen
  - Kerckhoff Klinik Forschungsgesellschaft, Bad Nauheim
  - Charité Campus Mitte, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Asklepios Klinik St. Georg, Hamburg
  - Universität Leipzig Herzzentrum, Leipzig
  - Medizinische Universitätsklinik Tübingen, Tübingen
- Netherlands (3):
  - Medisch Centrum Alkmaar, Alkmaar
  - Rijnland Ziekenhuis, Leiderdorp
  - UMC Maastricht, Maastricht
- Russia (2):
  - Scientific Research Institute of Circulation Pathology, Novosibirsk
  - Almazov Federal Heart, Blood & Endocrinolgoy Centre, Saint Petersburg
- Slovakia (2):
  - SsUSCH Baska Bystrica, Banská Bystrica
  - NUSCH Bratislava a.s., Bratislava

REFERENCES:
- [Background] Nergardh A, Frick M. Perceived heart rhythm in relation to ECG findings after direct current cardioversion of atrial fibrillation. Heart. 2006 Sep;92(9):1244-7. doi: 10.1136/hrt.2005.082156. Epub 2006 Mar 17. PMID 16547207
- [Background] Hindricks G, Piorkowski C, Tanner H, Kobza R, Gerds-Li JH, Carbucicchio C, Kottkamp H. Perception of atrial fibrillation before and after radiofrequency catheter ablation: relevance of asymptomatic arrhythmia recurrence. Circulation. 2005 Jul 19;112(3):307-13. doi: 10.1161/CIRCULATIONAHA.104.518837. Epub 2005 Jul 11. PMID 16009793
- [Background] Kimman GJ, Theuns DA, Janse PA, Rivero-Ayerza M, Scholten MF, Szili-Torok T, Jordaens LJ. One-year follow-up in a prospective, randomized study comparing radiofrequency and cryoablation of arrhythmias in Koch's triangle: clinical symptoms and event recording. Europace. 2006 Aug;8(8):592-5. doi: 10.1093/europace/eul051. Epub 2006 Jun 27. PMID 16803840
- [Background] Senatore G, Stabile G, Bertaglia E, Donnici G, De Simone A, Zoppo F, Turco P, Pascotto P, Fazzari M. Role of transtelephonic electrocardiographic monitoring in detecting short-term arrhythmia recurrences after radiofrequency ablation in patients with atrial fibrillation. J Am Coll Cardiol. 2005 Mar 15;45(6):873-6. doi: 10.1016/j.jacc.2004.11.050. PMID 15766823
- [Background] Patten M, Maas R, Karim A, Muller HW, Simonovsky R, Meinertz T. Event-recorder monitoring in the diagnosis of atrial fibrillation in symptomatic patients: subanalysis of the SOPAT trial. J Cardiovasc Electrophysiol. 2006 Nov;17(11):1216-20. doi: 10.1111/j.1540-8167.2006.00609.x. Epub 2006 Sep 20. PMID 16987384
- [Background] Fetsch T, Bauer P, Engberding R, Koch HP, Lukl J, Meinertz T, Oeff M, Seipel L, Trappe HJ, Treese N, Breithardt G; Prevention of Atrial Fibrillation after Cardioversion Investigators. Prevention of atrial fibrillation after cardioversion: results of the PAFAC trial. Eur Heart J. 2004 Aug;25(16):1385-94. doi: 10.1016/j.ehj.2004.04.015. PMID 15302102
- [Background] Kottkamp H, Tanner H, Kobza R, Schirdewahn P, Dorszewski A, Gerds-Li JH, Carbucicchio C, Piorkowski C, Hindricks G. Time courses and quantitative analysis of atrial fibrillation episode number and duration after circular plus linear left atrial lesions: trigger elimination or substrate modification: early or delayed cure? J Am Coll Cardiol. 2004 Aug 18;44(4):869-77. doi: 10.1016/j.jacc.2004.04.049. PMID 15312874
- [Background] Israel CW, Gronefeld G, Ehrlich JR, Li YG, Hohnloser SH. Long-term risk of recurrent atrial fibrillation as documented by an implantable monitoring device: implications for optimal patient care. J Am Coll Cardiol. 2004 Jan 7;43(1):47-52. doi: 10.1016/j.jacc.2003.08.027. PMID 14715182
- [Background] Strickberger SA, Ip J, Saksena S, Curry K, Bahnson TD, Ziegler PD. Relationship between atrial tachyarrhythmias and symptoms. Heart Rhythm. 2005 Feb;2(2):125-31. doi: 10.1016/j.hrthm.2004.10.042. PMID 15851283
- [Background] Ziegler PD, Koehler JL, Mehra R. Comparison of continuous versus intermittent monitoring of atrial arrhythmias. Heart Rhythm. 2006 Dec;3(12):1445-52. doi: 10.1016/j.hrthm.2006.07.030. Epub 2006 Aug 3. PMID 17161787
- [Background] Israel CW, Neubauer H, Olbrich HG, Hartung W, Treusch S, Hohnloser SH; BEATS Study Investigators. Incidence of atrial tachyarrhythmias in pacemaker patients: results from the Balanced Evaluation of Atrial Tachyarrhythmias in Stimulated patients (BEATS) study. Pacing Clin Electrophysiol. 2006 Jun;29(6):582-8. doi: 10.1111/j.1540-8159.2006.00405.x. PMID 16784423
- [Background] Joshi AK, Kowey PR, Prystowsky EN, Benditt DG, Cannom DS, Pratt CM, McNamara A, Sangrigoli RM. First experience with a Mobile Cardiac Outpatient Telemetry (MCOT) system for the diagnosis and management of cardiac arrhythmia. Am J Cardiol. 2005 Apr 1;95(7):878-81. doi: 10.1016/j.amjcard.2004.12.015. PMID 15781022
- [Background] Vasamreddy CR, Dalal D, Dong J, Cheng A, Spragg D, Lamiy SZ, Meininger G, Henrikson CA, Marine JE, Berger R, Calkins H. Symptomatic and asymptomatic atrial fibrillation in patients undergoing radiofrequency catheter ablation. J Cardiovasc Electrophysiol. 2006 Feb;17(2):134-9. doi: 10.1111/j.1540-8167.2006.00359.x. PMID 16533249
- [Derived] Hindricks G, Pokushalov E, Urban L, Taborsky M, Kuck KH, Lebedev D, Rieger G, Purerfellner H; XPECT Trial Investigators. Performance of a new leadless implantable cardiac monitor in detecting and quantifying atrial fibrillation: Results of the XPECT trial. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):141-7. doi: 10.1161/CIRCEP.109.877852. Epub 2010 Feb 16. PMID 20160169